CLINICAL TRIAL: NCT05006352
Title: A Phase 1b, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study, Followed by an Open-Label Extension, to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of DNL343 in Participants With Amyotrophic Lateral Sclerosis
Brief Title: A Study to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of DNL343 in Participants With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-F-0003; 2021-001766-37 (EudraCT Number)
Record Dates: First submitted 2021-08-07; First posted 2021-08-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DNL343 (High Dose) (Experimental)
  Interventions: Drug: DNL343
- DNL343 (Low Dose) (Experimental)
  Interventions: Drug: DNL343
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL343 — Oral repeating dose
  Arms: DNL343 (High Dose); DNL343 (Low Dose)
Drug: Placebo — Oral repeating dose
  Arms: Placebo

SUMMARY:
This is a Phase 1b, multicenter, randomized, placebo-controlled, double-blind study of 28 days, followed by an 18-month open-label extension, designed to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of DNL343 in participants with amyotrophic lateral sclerosis (ALS)

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of sporadic or familial ALS
* ≤ 4 years since ALS symptom onset
* Stable doses of approved ALS treatments (riluzole and/or edaravone) for at least 2 months prior to screening
* Participants must be able to swallow the study intervention
* Vital capacity >50% predicted at screening
* Women must have been surgically sterilized, be postmenopausal, or for participants of childbearing potential, must not be pregnant, and both the participant and the male partner must use highly effective contraception
* Men, and sex partner if a woman of childbearing potential, must use highly effective contraception

Key Exclusion Criteria:

* Any history of unstable or poorly controlled psychiatric, endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematologic, immunologic, or allergic disease, or other major disorders
* Positive serum pregnancy test or currently lactating or breastfeeding
* History of malignancy within 5 years
* History of clinically significant neurologic disorders other than ALS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) throughout the double-blind period | 28 Days

SECONDARY OUTCOMES:
PK parameter: Maximum concentration (Cmax) of DNL343 in plasma | 19 months
PK parameter: Time to reach maximum concentration (tmax) of DNL343 in plasma | 19 months
PK parameter: Trough concentration (Ctrough) of DNL343 in plasma | 19 months
PK parameter: Area under the concentration-time curve from time zero to 24 hours (AUC24) of DNL343 in plasma | 19 months
Cerebrospinal fluid-to-plasma concentration ratio of DNL343 following multiple oral doses | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Linus Sun, MD, PhD, Study Director — Denali Therapeutics Inc.
Locations (7):
- United States (6):
  - HonorHealth, Scottsdale, Arizona
  - University of California at San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - PPD Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Atrium Health Neurosciences Institute, Charlotte, North Carolina
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No